CLINICAL TRIAL: NCT00139113
Title: Immunogenicity Study of an Inactivated Hepatitis A Vaccine in Infants and Young Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Alaska Native Medical Center (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-NCID-1358; U50/CCU022279
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis A
Keywords: hepatitis A; hepatitis A vaccine
MeSH Terms: conditions — Hepatitis A; Hepatitis | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- HAVRIX 6 and 12 mos; mother antibody pos (Experimental): HAVRIX administered to infants born to anti-HAV positive mothers at ages 6 and 12 months
  Interventions: Biological: hepatitis A vaccine
- HAVRIX age 6, 12 mos; mom antibody neg (Active Comparator): HAVRIX administered to infants born to anti-HAV negative mothers at ages 6 and 12 months
  Interventions: Biological: hepatitis A vaccine
- HAVRIX ages 12, 15 mos; mom antibody + (Experimental): HAVRIX administered to infants born to anti-HAV positive mothers at ages 12 and 15 months
  Interventions: Biological: hepatitis A vaccine
- HAVRIX ages 12, 15 mos; mom antibody- (Active Comparator): HAVRIX administered to infants born to anti-HAV negative mothers at ages 12 and 15 months
  Interventions: Biological: hepatitis A vaccine
- HAVRIX ages 15,21 mos; mom antibody + (Experimental): HAVRIX administered to infants born to anti-HAV positive mothers at ages 15 and 21 months
  Interventions: Biological: hepatitis A vaccine
- HAVRIX ages 15,21 mos; mom antibody - (Active Comparator): HAVRIX administered to infants born to anti-HAV negative mothers at ages 15 and 21 months
  Interventions: Biological: hepatitis A vaccine

INTERVENTIONS:
Biological: hepatitis A vaccine — 2 doses of inactivated hepatitis A vaccine manufactured by GSK in licensed pediatric formulation of 720 EL. U. per dose given on 3 different schedules: aged 6 and 12 months, 12 and 18 months, and 15 and 21 months. Within each group, subjects were randomized to achieve a relatively equal number of children born to anti-HAV positive and anti-HAV negative mothers.
  Other Names: HAVRIX

SUMMARY:
Infants born to immune mothers and therefore having passively-transferred maternal antibody (PMA) to hepatitis A virus (HAV) have a blunted immune response to hepatitis A vaccine. We compared the immunogenicity of hepatitis A vaccine among infants with and without PMA, vaccinated on different schedules. We found that when vaccination is begun at or after 12 months of age, there was no difference in the immune response to the vaccine between infants born to immune vs. susceptible mothers.

DETAILED DESCRIPTION:
Background: Infants with passively-transferred maternal antibody (PMA) to hepatitis A virus (HAV) have a blunted immune response to hepatitis A vaccine. We compared the immunogenicity of hepatitis A vaccine among infants with and without PMA, vaccinated on different schedules.

Methods: Infants were randomized to one of three groups, each receiving two doses of 720 EL.U. of hepatitis A vaccine (HAVRIX, Glaxo SmithKline) according to the following schedules: Group 1 at ages 6 and 12 months; Group 2 at ages 12 and 18 months; Group 3 at ages 15 and 21 months. We determined antibody to HAV (anti-HAV) status of mothers at the time of delivery, and measured infants' anti-HAV concentrations at the time of the first vaccine dose (baseline), and at 1, 7 and 12 months thereafter. Anti-HAV concentrations > 33 milli-International Units/milliliter (mIU/mL) were considered protective. We monitored adverse reactions using diary cards and chart reviews.

Results: A total of 239 infants were enrolled, including 134 born to anti-HAV negative mothers (Groups 1N, 2N, 3N) and 105 born to anti-HAV positive mothers (Groups 1P, 2P, 3P).

At month 12, 6 months after the second vaccine dose, the difference in GMC between Groups 1P and 1N was the only statistically significant difference within groups (p<0.05). There were no statistically significant differences in GMC among groups of infants born to anti-HAV negative mothers ("N" groups), but the difference between Group 1P and Group 3P infants was significant (p < 0.05). No serious adverse reactions related to vaccination were detected.

Conclusions: Hepatitis A vaccine is immunogenic among infants born to anti-HAV negative mothers, and among those born to anti-HAV positive mothers and vaccinated beginning as young as 12 months old. The persistence of PMA for at least six months among the majority of infants born to anti-HAV positive mothers results in lower seroconversion rates and GMC's.

ELIGIBILITY:
Inclusion Criteria:term infant with normal growth and development, considered to be healthy at age 6 months; written informed consent by parent/guardian -

Exclusion Criteria:received or expected to receive immune globulin or blood/blood products while enrolled; received or expected to receive immunosuppressive therapy within 30 days of vaccination or has immune deficiency; currently enrolled in another vaccine trial; progressive or unstable neurological disorder

-

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 248 (Actual)
Dates: Start 1996-09; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
concentration of antibody to hepatitis A virus | baseline and 1, 7, and 12 months post vax
  Sera obtained at time of first hepatitis A vaccine dose (baseline) and 1, 7, and 12 months thereafter

SECONDARY OUTCOMES:
reported side effects and adverse events | day of vaccination and 3 days thereafter
  at time of each vaccine dose, parent was given a diary card on which to record systemic and injection site signs and symptoms observed on day of vaccination and subsequent 3 days.
antibodies to routine childhood vaccinations | age 13 months
  in a sample of study subjects from each group, blood drawn at age 13 months was tested for response to routine vaccinations.

CONTACTS AND LOCATIONS:
Overall Officials: Brian McMahon, Principal Investigator — Alaska Native Medical Center
Locations (2):
- United States (2):
  - Anchorage Neighborhood Health Center, Anchorage, Alaska
  - Alaska Native Medical Center, Anchorage, Alaska

REFERENCES:
- [Result] Bell BP, Negus S, Fiore AE, Plotnik J, Dhotre KB, Williams J, Shapiro CN, McMahon BJ. Immunogenicity of an inactivated hepatitis A vaccine in infants and young children. Pediatr Infect Dis J. 2007 Feb;26(2):116-22. doi: 10.1097/01.inf.0000253253.85640.cc. PMID 17259872